CLINICAL TRIAL: NCT00313144
Title: ARALAST alpha1-proteinase Inhibitor (α1-PI) Surveillance Study
Brief Title: Aralast alpha1-proteinase Inhibitor Surveillance Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early due to Aralast being phased out of the market.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 450501
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARALAST Alpha1-Proteinase Inhibitor — Weekly ARALAST infusions for 2 years, dose and mode of administration as prescribed by the physician

SUMMARY:
The primary objectives of this Phase 4, open label, prospective U.S. surveillance study are to evaluate the health outcomes of Alpha 1-Antitrypsin (AAT)-deficient subjects who are initiating treatment with ARALAST on patient-related outcomes (PRO), i.e., health-related quality of life (HRQoL), healthcare resource utilization (HCRU), and various laboratory analyses to evaluate the safety of long-term administration of ARALAST.

Up to 120 subjects will be enrolled and assessed for HRQoL and HCRU at baseline and every 6-months thereafter, for 2 years. A subset of subjects will be enrolled into the blood draw portion of the study, which will also include assessments of antibodies to ARALAST, and chemistry panel. Subjects will be treated according to the prescribing (attending) physician's instructions based on the prescribing information given in the ARALAST package insert.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Diagnosis of AAT deficiency associated emphysema
* Active prescription for augmentation therapy with ARALAST
* On service with Coram (a speciality pharmacy provider)
* Signed and dated informed consent

Exclusion Criteria:

* Clinically significant medical (other than COPD), psychiatric, or cognitive illness that, in the opinion of Coram or the sponsor or the investigator, may compromise subject safety or compliance (such as end stage renal or hepatic or heart disease, or metastatic cancer or any difficulty in communicating over the telephone lines)
* Previous treatment with ARALAST (i.e. subjects who had previously received and then discontinued ARALAST augmentation therapy and are now restarting ARALAST will be excluded from the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-06-09 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Adupa Rao, MD, San Marino, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a surveillance study conducted by Coram, Inc., in locations throughout the United States, and supervised by Baxter. Enrollment began in June 2006 and the study was terminated early, in December 2008, due to Aralast being phased out of the market.
Pre-assignment Details: 127 participants enrolled in the study, of these 126 participated in the health related quality of life (HRQoL) and healthcare resource utilization (HCRU) portion, 61 consented to the blood draw portion, and 66 only consented to the Quality of Life portion
Groups:
- Overall Study: Participants were treated with ARALAST according to dose and frequency of infusions recommended by their physician.
Period: Overall Study
Arm/Group | Overall Study
Started | 127
Completed | 17
Not Completed | 110
Not completed — Discontinue Aralast ≥4 consecutive doses | 12
Not completed — Death | 7
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 4
Not completed — Terminated by sponsor/ homecare provider | 4
Not completed — Physician Decision | 4
Not completed — Adverse event - transient | 5
Not completed — Liver transplant | 1
Not completed — Insurance (homecare provider) change | 1
Not completed — Change to different product | 1
Not completed — Due to termination of the study | 66

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 127
Age, Continuous [Median (Full Range); unit: years] | 52.3 [21.2 to 84.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127
Health Related Quality of Life (HRQoL): Baseline Assessment SF-36 Health Domain Scores (n=126) [Mean (Standard Deviation); unit: Scores on a scale] — The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary score (PCS)=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary score (MCS)=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score.
  Scores on a scale
    Physical Functioning (PF) | 31.612 (11.678)
    Role Limitation Due to Physical Health (RP) | 37.281 (11.871)
    Bodily Pain (BP) | 46.368 (11.116)
    General Health (GH) | 37.351 (10.120)
    Vitality (VT) | 42.279 (11.209)
    Social Functioning (SF) | 41.699 (14.069)
    Role Limitation Due to Emotional Problems (RE) | 48.474 (10.687)
    Mental Health (MH) | 47.326 (11.358)
    Physical Component Score (PCS) | 34.150 (11.263)
    Mental Component Score (MCS) | 50.340 (11.897)

OUTCOME MEASURES:

1. Primary Outcome: HRQoL 'Physical Functioning (PF)' From Baseline to ≤6 Months
Description: Change in quality of life survey response as measured using the SF-36 questionnaire. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores. The data transformation process was based on: Ware et al. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: Quality Metric Incorporated; 2000.
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 31.958 (11.291) | 33.129 (11.527)

2. Primary Outcome: HRQoL 'Role Limitation Due to Physical Health (RP)' From Baseline to ≤6 Months
Description: Change in quality of life survey response as measured using the SF-36 questionnaire. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores. The data transformation process was based on Ware et al. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: Quality Metric Incorporated; 2000.
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 37.631 (11.819) | 38.139 (11.338)

3. Primary Outcome: HRQoL 'Bodily Pain (BP)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 46.474 (10.895) | 48.950 (11.579)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.044, Paired t-test

4. Primary Outcome: HRQoL 'General Health (GH)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 37.365 (10.038) | 38.737 (10.490)

5. Primary Outcome: HRQoL 'Vitality (VT)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 42.578 (11.164) | 45.081 (10.916)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.009, Paired t-test

6. Primary Outcome: HRQoL 'Social Functioning (SF)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 42.340 (14.060) | 45.581 (12.780)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.005, Paired t-test

7. Primary Outcome: HRQoL 'Role Limitation Due to Emotional Problems (RE)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 48.361 (10.972) | 47.921 (10.855)

8. Primary Outcome: HRQoL 'Mental Health (MH)' From Baseline to ≤6 Months
Description: as for outcome 2
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 47.457 (10.711) | 50.007 (9.480)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.006, Paired t-test

9. Primary Outcome: HRQoL 'Physical Component Score (PCS)' From Baseline to ≤6 Months
Description: SF-36 scores for baseline (screening) versus the period from baseline to ≤6 Months. The PCS is a summary scale of the dimensions physical functioning, role physical, bodily pain, and general health. The component score is normalized to a standard population. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores.
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 34.453 (10.957) | 35.826 (10.881)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.044, Paired t-test

10. Primary Outcome: HRQoL 'Mental Component Score (MCS)' From Baseline to ≤6 Months
Description: SF-36 scores for baseline (screening) versus the period from baseline to ≤6 Months. The MCS is a summary scale of the dimensions vitality, social functioning, role emotional, and mental health Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores.
Time Frame: Screening to ≤ 6 Months
Population: Participants with baseline and participating during the period from baseline to ≤6 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months
Number analyzed (Participants) | 106 | 106
Scores on a scale | 50.464 (11.713) | 52.378 (10.639)
Statistical Analysis 1: Comparison: Baseline vs Baseline to ≤6 Months; Test type: Superiority or Other; p = 0.046, Paired t-test

11. Primary Outcome: HRQoL For: PF, RP, BP, GH, VT, SF, RE, MH, PCS, and MCS: Baseline, Baseline to ≤6 Months, and >6 Months to ≤12 Months
Description: SF-36 Scores- baseline thru 12 months, where data was available. Change in quality of life survey response as measured using the SF-36 questionnaire. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores. The Data transformation process was based on: Ware et al. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: Quality Metric Incorporated; 2000.
Time Frame: Baseline to 12 months
Population: Participants with baseline and participating during the period from baseline to ≤12 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months
Number analyzed (Participants) | 65 | 65 | 65
Scores on a scale
  Physical Functioning (PF) | 34.822 (11.173) | 35.632 (11.251) | 34.143 (11.914)
  Role Limitation Due to Physical Health (RP) | 40.539 (11.627) | 39.484 (11.615) | 38.542 (13.061)
  Bodily Pain (BP) | 47.203 (11.375) | 50.227 (11.267) | 47.788 (13.139)
  General Health (GH) | 38.853 (10.197) | 39.990 (10.013) | 40.026 (11.720)
  Vitality (VT) | 44.646 (11.546) | 45.703 (11.516) | 44.742 (11.058)
  Social Functioning (SF) | 44.683 (13.864) | 47.200 (11.799) | 43.927 (14.384)
  Role Limitation Due to Emotional Problems (RE) | 48.403 (11.214) | 48.583 (10.590) | 48.942 (12.011)
  Mental Health (MH) | 47.365 (11.040) | 50.311 (8.962) | 49.488 (11.705)
  Physical Component Score (PCS) | 37.346 (10.906) | 37.890 (10.499) | 36.272 (11.238)
  Mental Component Score (MCS) | 50.442 (11.896) | 52.508 (10.354) | 51.854 (12.088)

12. Primary Outcome: HRQoL for PF, RP, BP, GH, VT, SF, RE, MH, PCS, and MCS Scores: Baseline, Baseline to ≤6 Months, >6 Months to ≤12 Months, and >12 Months to ≤18 Months
Description: as for outcome 11
Time Frame: Baseline to 12 months
Population: Participants with baseline and participating during the period from baseline to ≤18 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months
Number analyzed (Participants) | 47 | 47 | 47 | 47
Scores on a scale
  Physical Functioning (PF) | 34.197 (11.375) | 34.958 (11.048) | 33.301 (11.764) | 33.839 (12.546)
  Role Limitation Due to Physical Health (RP) | 40.492 (12.310) | 39.033 (11.686) | 37.887 (12.964) | 40.336 (12.324)
  Bodily Pain (BP) | 47.525 (12.023) | 50.726 (10.942) | 48.990 (13.177) | 50.537 (11.789)
  General Health (GH) | 38.684 (10.164) | 39.718 (9.697) | 39.475 (11.435) | 39.586 (10.848)
  Vitality (VT) | 45.714 (11.843) | 46.245 (10.807) | 45.249 (11.002) | 45.648 (10.901)
  Social Functioning (SF) | 45.825 (14.089) | 47.218 (11.665) | 44.781 (14.110) | 45.013 (14.127)
  Role Limitation Due to Emotional Problems (RE) | 49.014 (11.497) | 48.187 (11.158) | 48.022 (13.331) | 47.360 (11.930)
  Mental Health (MH) | 48.390 (11.740) | 50.187 (9.347) | 49.229 (12.562) | 48.569 (11.902)
  Physical Component Score (PCS) | 36.803 (11.105) | 37.655 (10.609) | 36.171 (10.848) | 38.060 (11.450)
  Mental Component Score (MCS) | 51.885 (12.215) | 52.575 (10.846) | 51.843 (13.323) | 50.814 (12.729)

13. Primary Outcome: HRQoL for PF, RP, BP, GH, VT, SF, RE, MH, PCS, and MCS Scores: Baseline, Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months
Description: SF-36 Scores- baseline thru 24 months, where data was available. Change in quality of life survey response as measured using the SF-36 questionnaire. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores. The Data transformation process was based on: Ware et al. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: Quality Metric Incorporated; 2000.
Time Frame: Baseline to 24 months
Population: Participants with baseline and participating during the period from baseline to ≤24 months data for HRQoL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
Scores on a scale
  Physical Functioning (PF) | 36.489 (11.174) | 35.988 (10.874) | 34.585 (12.241) | 35.487 (12.782) | 33.883 (12.836)
  Role Limitation Due to Physical Health (RP) | 43.092 (13.267) | 42.509 (11.390) | 40.643 (13.245) | 42.276 (11.577) | 41.576 (12.841)
  Bodily Pain (BP) | 52.036 (13.330) | 53.988 (11.695) | 52.559 (14.045) | 56.041 (10.951) | 51.674 (12.214)
  General Health (GH) | 38.452 (11.496) | 40.744 (10.222) | 39.632 (11.720) | 40.245 (11.852) | 38.293 (11.171)
  Vitality (VT) | 47.036 (11.949) | 48.969 (10.116) | 49.118 (10.187) | 47.036 (9.797) | 47.631 (10.705)
  Social Functioning (SF) | 46.980 (16.418) | 48.538 (12.026) | 44.123 (14.361) | 46.980 (13.756) | 48.019 (15.181)
  Role Limitation Due to Emotional Problems (RE) | 49.215 (14.077) | 49.400 (12.002) | 49.770 (12.984) | 49.770 (12.142) | 49.030 (12.348)
  Mental Health (MH) | 48.801 (13.404) | 50.007 (10.686) | 50.812 (13.626) | 49.471 (12.581) | 50.276 (13.084)
  Physical Component Score (PCS) | 39.963 (11.722) | 40.480 (11.113) | 38.287 (12.037) | 40.716 (10.711) | 37.890 (12.785)
  Mental Component Score (MCS) | 51.510 (14.484) | 53.011 (12.441) | 53.120 (13.910) | 51.990 (12.726) | 53.389 (15.119)

14. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Frequency of Emergency Room (ER) Visits'
Description: Number of participants with indicated number of ER visits (0, 1, 2, 3, ≥4 ER visits per participant) during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: Baseline to 24 Months
Population: Participants with data available during each window period
Measure: Number; unit: Participants
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 106 | 65 | 47 | 21
Participants
  0 ER visits | 84 | 49 | 41 | 19
  1 ER visits | 16 | 14 | 5 | 2
  2 ER visits | 5 | 2 | 1 | 0
  3 ER visits | 1 | 0 | 0 | 0
  ≥4 ER visits | 0 | 0 | 0 | 0

15. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Mean Number of Emergency Room (ER) Visits'
Description: Mean number of ER visits one year prior to baseline/screening, and during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: One year prior to baseline to 24 months post-baseline
Population: Participants with data available during each window period
Measure: Mean (Standard Deviation); unit: ER visits per time period
Arm/Group | Year Prior to Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 126 | 106 | 65 | 47 | 21
ER visits per time period | 0.85 (1.492) | 0.274 (0.594) | 0.28 (0.516) | 0.15 (0.416) | 0.10 (0.301)

16. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Frequency of Hospitalizations'
Description: Number of participants with indicated number of hospitalizations during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: Baseline to 24 Months
Population: Participants with data available during each window period
Measure: Number; unit: Participants
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 106 | 65 | 47 | 21
Participants
  0 Hospitalizations | 86 | 58 | 45 | 20
  1 Hospitalizations | 17 | 6 | 1 | 1
  2 Hospitalizations | 2 | 1 | 1 | 0
  3 Hospitalizations | 1 | 0 | 0 | 0
  ≥4 Hospitalizations | 0 | 0 | 0 | 0

17. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Mean Length of Stay (LOS) in Hospital'
Description: Mean LOS during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: Baseline to 24 months
Population: Participants with data available during each window period
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 106 | 65 | 47 | 21
Days | 0.8585 (2.29467) | 0.6462 (2.68346) | 0.25532 (1.374742) | 1.1905 (5.45545)

18. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Number of Participants Taking Antibiotics'
Description: Number of participants taking antibiotics one year prior to baseline/screening, and during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: One year prior to baseline to 24 months post-baseline
Population: Participants with data available during each window period
Measure: Number; unit: Participants
Arm/Group | Year Prior to Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 127 | 106 | 65 | 47 | 21
Participants | 90 | 58 | 37 | 25 | 8

19. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Number of Antibiotic Courses'
Description: Number of antibiotic courses (i.e. number of antibiotic prescriptions) one year prior to baseline/screening, and during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: One year prior to baseline to 24 months post-baseline
Population: Participants with data available during each window period
Measure: Mean (Standard Deviation); unit: Antibiotic courses
Arm/Group | Year Prior to Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 126 | 106 | 65 | 47 | 21
Antibiotic courses
  All antibiotic courses (oral and I.V.) | 2.3095 (2.84384) | 0.9906 (1.27612) | 0.9231 (1.07975) | 0.9787 (1.40634) | 0.7143 (1.18924)
  Oral antibiotic courses | 1.8571 (2.39571) | 0.8679 (1.08738) | 0.8154 (0.96651) | 0.8936 (1.25515) | 0.6667 (1.19722)
  I.V. antibiotic courses | 0.4603 (1.08555) | 0.1038 (0.36330) | 0.1077 (0.35895) | 0.0851 (0.28206) | 0.0476 (0.21822)

20. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Number of Participants Receiving Steroid Pulse Courses'
Description: Number of participants receiving steroid pulse courses (i.e. number of steroid prescriptions) one year prior to baseline/screening, and during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: One year prior to baseline to 24 months post-baseline
Population: Participants with data available during each window period
Measure: Number; unit: Participants
Arm/Group | Year Prior to Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 127 | 106 | 65 | 47 | 21
Participants | 65 | 30 | 14 | 12 | 4

21. Secondary Outcome: Healthcare Resource Utilization (HCRU) 'Number of Steroid Pulse Courses'
Description: Number of steroid pulse courses (i.e. number of steroid prescriptions) one year prior to baseline/screening, and during each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: One year prior to baseline to 24 months post-baseline
Population: Participants with data available during each window period
Measure: Mean (Standard Deviation); unit: Steroid Pulse Courses
Arm/Group | Year Prior to Baseline | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 126 | 106 | 65 | 47 | 21
Steroid Pulse Courses
  All steroid pulse courses (oral and I.V.) | 1.4365 (2.51554) | 0.4340 (0.89463) | 0.4154 (1.07372) | 0.3404 (0.66844) | 0.2857 (0.71714)
  Oral steroid pulse courses | 1.0873 (2.13174) | 0.3585 (0.84164) | 0.3692 (1.03937) | 0.2766 (0.53981) | 0.2381 (0.70034)
  I.V. steroid pulse courses | 0.3492 (0.96596) | 0.0849 (0.28007) | 0.0462 (0.21145) | 0.0638 (0.24709) | 0.0476 (0.21822)

22. Secondary Outcome: Hepatic Chemistry Parameters: Change From Baseline/Screening
Description: Summary of changes in hepatic (total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase) parameters from screening/baseline through each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: Baseline to 24 months
Population: Subjects who participated in the blood draws with data available during each window period
Measure: Median (Full Range); unit: U/L
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 52 | 34 | 26 | 15
U/L
  Alkaline phosphatase | -1.00 [-39.0 to 33.0] | 1.50 [-68.0 to 35.0] | -5.50 [-70.0 to 21.0] | 0.00 [-61.0 to 13.0]
  ALT | 0.00 [-21.0 to 27.0] | 2.50 [-19.0 to 26.0] | 2.00 [-21.0 to 35.0] | 2.00 [-27.0 to 11.0]
  AST | 1.00 [-25.0 to 22.0] | 0.00 [-23.0 to 9.0] | 1.00 [-17.0 to 27.0] | 0.00 [-10.0 to 7.0]

23. Secondary Outcome: Renal and Hepatic Chemistry Parameters: Change From Baseline/Screening
Description: Summary of changes in hepatic (total bilirubin) and renal (Blood urea nitrogen (BUN), creatinine) parameters from screening/baseline through each window period (Baseline to ≤6 Months, >6 Months to ≤12 Months, >12 Months to ≤18 Months, and >18 Months to ≤24 Months)
Time Frame: Baseline to 24 months
Population: Subjects who participated in the blood draws with data available during each window period
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 52 | 34 | 26 | 15
mg/dL
  Creatinine | 0.02 [-0.2 to 0.6] | 0.01 [-0.1 to 0.3] | 0.04 [-0.2 to 0.2] | 0.00 [-0.2 to 0.2]
  Total bilirubin | 0.00 [-0.7 to 0.6] | 0.00 [-0.5 to 0.5] | 0.00 [-0.3 to 0.6] | 0.00 [-0.5 to 0.5]
  BUN | 0.65 [-7.7 to 9.8] | -0.15 [-9.2 to 10.7] | 1.50 [-8.4 to 7.7] | -0.50 [-4.3 to 9.0]

24. Secondary Outcome: ARALAST Antibody Titers: Participants With at Least 2-Dilution Step Increases From Screening
Description: All IgG and IgM titers at screening were ≤ 4. A 2-dilution step increase was defined as follows: • The titer at each 6-month visit must be ≥ 4 when the screening titer = 0 • Each 6-month visit titer / screening titer should be ≥ 4. 6 month window periods are: baseline to ≤6 months, >6 months to ≤12 months, >12 months to ≤18 months, and >18 months to ≤24 months
Time Frame: Baseline to 24 Months
Population: Subjects who participated in the blood draws with data available during each window period
Measure: Number; unit: Participants
Arm/Group | Baseline to ≤6 Months | >6 Months to ≤12 Months | >12 Months to ≤18 Months | >18 Months to ≤24 Months
Number analyzed (Participants) | 52 | 34 | 26 | 15
Participants
  IgG | 2 | 0 | 0 | 0
  IgM | 2 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (2 years, 7 months)
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 39/127
Other Adverse Events (participants affected / at risk) | 97/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=127)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Colon gangrene (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Hernia (General disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Pseudomonas infection (Infections and infestations) | 1 (2)
Respiratory tract infection (Infections and infestations) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Disorientation (Nervous system disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=127)
Diarrhea (Gastrointestinal disorders) | 7 (21)
Fatigue (General disorders) | 15 (123)
Infusion related reaction (General disorders) | 9 (13)
Hypersensitivity (Immune system disorders) | 13 (28)
Influenza (Infections and infestations) | 7 (27)
Lower respiratory tract infection (Infections and infestations) | 24 (35)
Oral fungal infection (Infections and infestations) | 10 (18)
Respiratory tract infection (Infections and infestations) | 33 (66)
Upper respiratory tract infection (Infections and infestations) | 28 (45)
Headache (Nervous system disorders) | 23 (98)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 (33)
Elective procedure (Surgical and medical procedures) | 8 (9)
Poor venous access (Vascular disorders) | 8 (10)

LIMITATIONS AND CAVEATS:
Study was terminated early due to Aralast being phased out of the market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. Baxter may require a review of results communications (e.g., for confidential information & intellectual property) ≥45 days prior to submission or communication for review and comment. Baxter reserves the right to remove all confidential information from all publications.